CLINICAL TRIAL: NCT00601029
Title: Rhabdomyolysis in Basic Training
Status: Completed | Type: Observational
Sponsor: Martin Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rodney S. Gonzalez, MD, Chief, Warrior Care, Martin Army Community Hospital
Other Study IDs: DDEAMC 07-25; USUHS G192FP; CIRO 2007522
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Exertional Rhabdomyolysis
Keywords: Exertional Rhabdomyolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and stored blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Winter Phase - Observational
- 2: Summer Phase - Observational

SUMMARY:
The purpose of this study is to:

1. develop a normative database for serum creatine kinase (CK) responses to basic military training (BMT);
2. determine the incidence of exertional rhabdomyolysis (ER) among a large cohort of recruits undergoing BMT;
3. assess the impact of climate on the incidence of ER during BMT;
4. determine the incidence of candidate genes that may be associated with an increased risk of ER.

DETAILED DESCRIPTION:
Based on our review of scientific information, we have identified several genetic varieties or polymorphisms that may be associated with an increased risk of muscle injury and/or heat illness. As part of our recruitment process we have provided you with this written study information, and will present to you a brief oral and PowerPoint presentation of the study design and schedule, and the time to address any questions not yet answered prior to issuing consent forms for those agreeing to participate.

Participation in this study is entirely voluntary; either agreeing or refusing to participate will have absolutely no effect on your status as a recruit or your standing in basic training. You will not be paid for your participation in this study. While your drill sergeant and company commander will be aware of all those who are participating in the study, this will occur only for scheduling purposes so that you and fellow participants can be excused for the 3 blood draws that will take place after basic physical training has begun. When you consent to participate in this study, you may place limitations on the use of your blood sample by selecting one of the options provided on the last page of the consent form. If at any point you decide not to continue in the study, detailed instructions for withdrawal are in the consent form.

Potential Risks: Participation in this study itself will not increase your risk of developing rhabdomyolysis. If you or any other participant should develop either rhabdomyolysis or very high CK levels, we will perform additional DNA analyses for certain conditions associated with exercise intolerance. Several of these are inherited muscle diseases that may not be diagnosed until adulthood and may only first become apparent after an episode of exercise intolerance. Diagnosis of any of these conditions is grounds for dismissal from the Army, but it is essential that you and your family be aware of these hereditary conditions if present.

Risks Associated With Genetic Analysis: There are certain additional risks that are uniquely associated with any study involving genetic testing. Using advanced genetic analysis, information about your DNA structure (genetic information) can help determine your risk of developing certain genetic diseases that run in families. This genetic information is unique to you and may indicate changes in your future health status or life expectancy, as well as possibly, that of your children and other relatives. Besides medical risks, genetic testing carries certain social risks. It can affect insurability, employability, personal family planning, family relationships, immigration status, instigate paternity lawsuits, and be associated with social stigmatization. Finding out that either you do or do not carry a gene associated with a serious illness can cause both significant stress and psychological harm.

Privacy and Confidentiality: All information provided, as part of this study will be confidential and protected to the fullest extent provided by law. Information and other records related to this study will be accessible to those persons directly involved in conducting this study and members of the Eisenhower Army Medical Center Institutional Review Committee (IRC), USUHS Research Department, and other governmental agencies, which provides oversight for protection of human research volunteers. All questionnaires, forms, and charts will be kept in a restricted-access, locked cabinet while not in use and blood samples will be stored in a restricted access, locked freezer at USUHS for up to five years, depending on how participants wish their blood to be used. After five years all remaining blood samples will be destroyed along with the code logbook. To enhance privacy of the information, all data will be entered into a database in which individual responses are not identified. After verification of the database information, all paper copies containing identifiers will be shredded.

You will not be informed of the general results of the study since this is a research study, but may review the literature for published results. However, if the results reveal that you have a mutation in any gene that indicates susceptibility to specific disorders (malignant hyperthermia, CPT II deficiency, McArdle's, AMP deaminase deficiency and MCAD deficiency), you will be informed; we will also inform your General Medical Officer (GMO). If you need a genetic counselor, we will arrange for this as well through your GMO. The genetic results that are not associated with dismissal from military service will not be released to anyone including you.

Complete confidentiality cannot be promised, particularly for military personnel, because information bearing on your health may be required to be reported to appropriate medical or command authorities.

Data Management: Data storage and analysis will be conducted on a desktop computer. The computer storing these data will be backed up daily and only the PI and the data manager will have access to the hard drive or discs. One copy of the disc will be maintained in a secure locked office. A copy of the data set will also be stored on one the of the USUHS servers by using a secure site, which is backed up daily.

Data files will be converted to SPSS™ datasets for processing and merging with other participant research data. For the written questionnaires and forms, the project will use a computer data management and analysis system composed of digital scanning technology with Teleform™. This technique minimizes data entry errors and cleans data files on an on-going basis. In addition, built-in range detection strategies will identify outliers that may represent errors. In brief, forms completed by participants will be scanned by an optical scanner and interpreted by Teleform™ Reader, which then checks for missing, illogical, and out-of-range values. The Reader also identifies data that have been (1) incorrectly completed, or (2) mistakenly marked, and (3) characters that do not satisfy the Reader's confidence level. Those that do not meet these parameters are held for manual review and correction. Correction is done with the Teleform™ Verifier. Once verification is complete, the data are exported to SPSS™ database software for statistical analysis. The database is programmed to check for illicit values and to calculate parameters derived from raw data.

Storage of Participant Samples: Your blood samples will be stored in appropriate conditions. All samples will be given a numerical code and stored without participant name or any other identifiers. This code will be entered into a logbook maintained by Dr. William Campbell or appropriate persons. All samples will be stored at the USUHS for 5 years unless otherwise instructed by the participant.

Use of Sample by Investigators: The protocol has specified the genes to be examined. However, over the course of the study, other candidate genes with identified polymorphisms may appear in the literature. If there is a clear justification for examining them for an association to rhabdomyolysis, we will carry out the analysis after contacting you and obtaining your permission. All of our analyses will relate specifically to the stated objectives and not unrelated research efforts. There will not be any secondary use of the samples obtained from the subjects since samples will not be shared with other investigators outside this study. The blood samples obtained from this research will not be used for any commercial purpose.

Withdrawal from Research: You have the right to withdraw from the study and have the option of withdrawing your blood sample(s) at any time. If you decide to stop your participation in the study, you need to contact the medical monitor and/or one of the members of the research team and inform any one of them of your decision. They will withdraw you from the study and no further blood samples, questionnaires or muscle exams will be performed. If your participation in this study is stopped before the end of the study, any information that has already been collected will be kept by the research team and included in study results. This information will be maintained for the duration of the study.

Participant Resource: Members of the study team will be available to answer questions from you at any time during the study, and in particular, during the three brief exams and blood draws while in the field. In addition, the medical monitor of the study, Dr. Michael Campbell, will also serve as the study ombudsman and be available as a resource to you or any study participant.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Basic Training at Ft. Benning
* Between the ages of 18 and 45
* Active Duty
* Able to speak and read English
* Held in inprocessing seven days or less

Exclusion Criteria:

* A no answer to any of the above inclusion criteria

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Military Basic Trainee at Ft. Benning undergoing Infantry Basic Training Male > 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Exertional Rhabdomyolysis | Day 0, 3, 7 and 14 of basic training

CONTACTS AND LOCATIONS:
Overall Officials: Rodney S Gonzalez, MD, Principal Investigator — Martin Army Community Hospital
Locations (1):
- Martin Army Community Hospital, Fort Benning, Georgia, United States